CLINICAL TRIAL: NCT03686319
Title: The Effect of Reflexology on Lactation and Postpartum Comfort for Cesarean-delivery
Brief Title: The Effect of Reflexology on Lactation and Postpartum Comfort for Cesarean-delivery Primiparous Mothers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Selcuk University (Other)
Responsible Party: Principal Investigator, seyhan Çankaya, Asistant Professor, Selcuk University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 99950669/53
Record Dates: First submitted 2018-09-24; First posted 2018-09-26 (Actual); Last update posted 2018-09-26 (Actual); Status verified 2018-09

CONDITIONS: Breastfeeding; Lactation Failure; Nursing Caries; Postpartum; Reflexology
MeSH Terms: conditions — Breast Feeding | interventions — Musculoskeletal Manipulations

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control groups (No Intervention): Primiparas appropriate for the criteria, admitted to the clinic due to CS and accepting to participate in the study were randomly placed into groups. Reflexology was performed in the intervention group mothers, and the questionnaires and scales were self-reportingly filled in by the lead researcher (SC).
  Different rooms were allocated for the participants in the intervention and control groups not to affect each other.
- "intervention" (foot reflexology) (Experimental): Reflexology was performed in those in the intervention group after CS on right foot for 10 min and left foot for 20 min as continuing 30-min seances three times per day every eight hours for three days. The procedure was started at mean 3rd hour after mothers became stable. Reflexology was performed for none of those in the control group.
  Interventions: Other: Reflexology

INTERVENTIONS:
Other: Reflexology — Reflexology: foot massage
  Arms: "intervention" (foot reflexology)

SUMMARY:
Immediately after cesarean birth, many women suffer from breastfeeding problems due to pain, fatigue, activity intolerance, anesthesia, and delayed onset of lactation. Because of these avoidable problems, the baby cannot get enough breast milk, and mothers' postpartum comfort decreases.

This study aimed to investigate the effect of reflexology on lactation and postpartum comfort in primiparas giving births through cesarean section.

DETAILED DESCRIPTION:
Methods: This randomized controlled trial was conducted with 100 women with first birth through cesarean section were investigated between May 2016 and May 2017. Expectant mothers were randomly included into an intervention and a control group. The intervention group consisted of mothers for whom reflexology was performed three times per day for 30 min every eight hours.

With face-to-face interviews, all participants were informed about the design, content and methods to be used in the study, and the sociodemographic data obtained self-reportingly from the primiparas were recorded. The data were collected between May 2016 and May 2017. In collecting the data related to primiparas and infants, a questionnaire structured by the researchers in light of literature was used, as well as The breastfeeding charting system (LATCH), The visual analogue scale (VAS) for signs of onset of lactation and The postpartum comfort questionnaire (PPCQ).

ELIGIBILITY:
Inclusion Criteria:

* primiparas delivering through CS,
* at the age of 18 and over,
* at ≤37 gestational weeks
* with one-fetus birth,
* with stable vital signs,
* those delivering under general anesthesia,
* except for CS and spinal/epidural anesthesia,
* with ability of communication in Turkish, and those accepting to participate into the study voluntarily.

Exclusion Criteria:

* primiparas with infectious diseases such as shingles, fungus, eczema, warts and callus in the intervention group,
* those with local infections like abscess,
* open lesion/wound, scar tissue, edema, hematoma, thrombophlebitis, deep vein thrombosis, coagulopathy, mass, varicosis, deformities on toes, recent fractures or dislocations, tearing of fascia and tendons,
* and with psychiatric disorders such as anxiety and depression, were excluded out of the study.

Ages: 18 Years to 41 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2016-05-01 (Actual); Primary Completion 2017-04-01 (Actual); Study Completion 2017-05-30 (Actual)

PRIMARY OUTCOMES:
The breastfeeding charting system (LATCH) | Change from The breastfeeding charting system (LATCH) scores at first, second and third days after cesarean.
  As nurses are more likely to use a subjective criterion as poor /fair/ well to document and assess breastfeeding, LATCH provides a systematic method to collect information about individual breastfeeding sessions. The system is scored between 0 and 5 to indicate the key components of breastfeeding. Each breastfeeding session is assessed in light of the total score. A total score lower than 10 means that mothers are to be supported (Yenal and Okumus, 2003; Demirhan, 1997; Jensen et al., 1995). The letters of the acronym LATCH designate separate areas of assessment: ''L'' for how well infants latch onto the breast, ''A'' for the amount of audible swallowing,''T'' for mothers' nipple type, ''C'' for mothers' level of comfort, ''H'' for the amount of support given for infants to hold the breast.
The visual analogue scale (VAS) for signs of onset of lactation | Change from The visual analogue scale (VAS) for signs of onset of lactation scores at first, second and third days after cesarean
  VAS was used to evaluate breast changes during the onset of lactation by mothers' self-reports, as in the study performed by Mauri et al. (2015). Initial signs of lactation were assessed as breast-tension, increase in breast-heat and breast-pain, and scored from 0 (no signs) to 10 (most powerful signs) (Mauri et al., 2015).
The postpartum comfort questionnaire (PPCQ) | At the end of 3rd day, The postpartum comfort questionnaire (PPCQ) was performed for all mothers.
  Constituted by Kolcaba in 1992, the General Comfort Scale (GCS) was adapted to Turkish by Kuguoglu and Karabacak in 2004 (Kuguoglu and Karabacak, 2008). Based on the Turkish version of GCS, the Postpartum Comfort Questionnaire (PPCQ) was developed by Karakaplan and Yildiz in 2010. Factor analyses were assigned to test the validity and reliability of GCS. The internal consistency in terms of reliability was tested, and the Cronbach's alpha was found as 0.78. PPCQ evaluates the physical, psychospiritual and sociocultural comfort of mothers after CS or vaginal delivery. These comfort areas also constitute the subdimensions of the scale. The scale using a 5-point Likert-type scoring includes 34 items, ranging from 5 (strongly agree) as the highest level of comfort to 1 (strongly disagree) as the lowest. Reverse coding is applied to the items with negative statements. The minimum and the maximum scores on the scale change between 34 and 170. The scores close to 170 indicate a high level of